CLINICAL TRIAL: NCT02600039
Title: The Short-term Effect of ELTGOL on Pulmonary Ventilation Valued Through Electrical Impedance Tomography in Cystic Fibrosis Patients: Randomized Crossover Study
Brief Title: The Short-term Effect of ELTGOL on Pulmonary Ventilation Valued Through Electrical Impedance Tomography in Cystic Fibrosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Amanda Silva Couto, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 37906314.3.0000.5208
Record Dates: First submitted 2015-10-29; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELTGOL (Experimental)
  Interventions: Other: ELTGOL; Device: Acapella
- Acapella (Active Comparator)
  Interventions: Other: ELTGOL; Device: Acapella

INTERVENTIONS:
Other: ELTGOL — Individuals will be placed in the lateral decubitus position and instructed to perform slow expirations with an open glottis through a nozzle attached to the mouth from the residual functional capacity to residual volume. Concurrently, a trained and subsequently positioned relative to the voluntary physical therapist will perform a manual compression of the abdominal region dependent and the rib cage to enhance contralateral lung deflation. This intervention is performed so that the time is homogeneous between each repetition interval of one minute between each set. To this end, three sets of ten repetitions will be performed on each lateral decubitus (left and right)
Device: Acapella — Participant should be comfortably seated and with his elbows on a table. The mouthpiece is attached properly to not allow leaks. The resistance load will be one in which the individual is able to maintain uninterrupted expiration of 3 seconds. Then the patient will be instructed to inhale slowly and deeply, with lung volumes between the residual volume and total lung capacity. The air exhaled by Acapella is directed toward an orifice which opens and closes periodically, promoting oscillations in the air stream throughout the expiratory phase. The expiration is always performed to the VR, and without performing the active contraction of the abdominal muscles. Still prompted an inspiratory pause of 2 seconds for the end of the inspiratory phase. This procedure will be performed in 4 sets of 5 minutes with interval of 1 minute between the series.

SUMMARY:
Cystic Fibrosis (CF) is the most common lethal autosomal recessive disease. Respiratory therapy is always recommended to the CF patient with pulmonary involvement and has differents techniques and devices, however, there is no consensus on the effectiveness of the techniques used, there is a need to determine the applicability of the therapeutic resources used. Therefore, the aim of the study is to determine the short-term effectiveness of ELTGOL on Average Electrical Impedance on the End of Expiration (MIEFE) pulmonary, assessed by Electrical Impedance Tomography (EIT) in individuals with CF through a clinical trial randomized crossover. Volunteers will be included with FC with moderate to severe lung disease with chest ≥ 74 cm that do not show: episode of pulmonary infectious exacerbations in the last four weeks or during the study period; cor pulmonale; facial deformity that causes air leakage; facial trauma and recent face or esophagus surgery; chest pain; hemoptysis in the last week; continued use of supplemental oxygen (> 8 hours / day); hemoptysis; hemodynamic instability and do not understand the use and command of the techniques used. The sample is selected by convenience from the database of individuals assisted data in Integrative Medicine Institute Professor Fernando Figueira (IMIP). The research will be developed in three phases, divided into three days with an interval of at least 48 hours between phases. The first day will undergo initial assessment and in the days following the intervention by day, ELTGOL or Acapella, in a randomized order.

ELIGIBILITY:
Inclusion Criteria: Volunteers with Cystic Fibrosis and lung disease with chest hemiperímetro ≥ 37 cm. Exclusion Criteria: Episode of pulmonary infectious exacerbations in the last four weeks or during the study period; cor pulmonale; facial deformity that causes air leakage; facial trauma and recent face or esophagus surgery; chest pain; hemoptysis in the last week; continued use of supplemental oxygen (> 8 hours / day); hemoptysis; hemodynamic instability and do not understand the use and command of the techniques used.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Average Electrical Impedance on the End-Expiration | up to 30 minutes

SECONDARY OUTCOMES:
Dyspnea assessed by the Borg scale | baseline, one minute and thirtieth minutes
Oxygen saturation assessed by oximeter | baseline, one minute and thirtieth minutes
Preferred technique assessed by an open question | up to 3 minutes
Adverse Effects associeted with ELTGOL and Acapella assessed by an open question | baseline, one minute and thirtieth minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil